CLINICAL TRIAL: NCT05687461
Title: Construction of a National Diagnosis and Treatment Quality Control Platform for Major Respiratory Diseases and Technical Promotion of Standardized Diagnosis and Treatment Programs
Brief Title: Construction of a National Diagnosis and Treatment Quality Control Platform for Major Respiratory Diseases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhenguo Zhai,MD,PhD, Chief physician, China-Japan Friendship Hospital
Other Study IDs: 12100000400014014Y
Record Dates: First submitted 2022-12-29; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Quality Control
Keywords: Quality Control; Respiratory Diseases
MeSH Terms: conditions — Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (2):
- People at high risk for VTE: Patients who are admitted to the hospital for acute medical illness or surgery operations.
  Interventions: Other: Build a national diagnosis and treatment quality control platform for major respiratory diseases
- People diagnosed with VTE: Patients who were clearly diagnosed with deep vein thrombosis or pulmonary thromboembolism.
  Interventions: Other: Build a national diagnosis and treatment quality control platform for major respiratory diseases

INTERVENTIONS:
Other: Build a national diagnosis and treatment quality control platform for major respiratory diseases — 1. Build a national diagnosis and treatment quality control platform for major respiratory diseases
  2. To master the incidence trend and diagnosis and treatment quality of major respiratory diseases
  3. Promotion of standardized diagnosis and treatment techniques for major respiratory diseases

SUMMARY:
1. Build a national diagnosis and treatment quality control platform for major respiratory diseases It will establish and improved a "National diagnosis and Treatment quality control Platform for major respiratory diseases", and form a three-level network of diagnosis and treatment quality control for major respiratory diseases with a three-level system structure of "national, provincial and hospital".
2. Promote standardized diagnosis and treatment techniques for major respiratory diseases Relying on the specialized disease collaboration group or innovative unit model, all-round and hierarchical precision training and teaching are carried out to popularize and promote standardized diagnosis and treatment technology schemes for major respiratory diseases, so as to achieve the homogenization of diagnosis and treatment level for major respiratory diseases.

DETAILED DESCRIPTION:
1. Build a national diagnosis and treatment quality control platform for major respiratory diseases Cooperate with the Medical Administration Administration of the National Health Commission, the Medical Administration Institute of the National Health Commission and the National Center for Respiratory Disease Medical Quality Control to integrate the existing diagnosis and treatment quality indicators and data from NCIS (National Medical Quality Management and Control Information Network) and HQMS (Hospital Quality Monitoring System), and determine the definition, data sources and collection rules of core quality control indicators. It has established and improved a "National diagnosis and Treatment quality control Platform for major respiratory diseases", and formed a three-level network of diagnosis and treatment quality control for major respiratory diseases with a three-level system structure of "national, provincial and hospital".
2. To master the incidence trend and diagnosis and treatment quality of major respiratory diseases Through the big data integration and analysis function of the "National Diagnosis and Treatment Quality Control Platform for Major Respiratory Diseases", the incidence trend and law of various major respiratory diseases are mastered. To understand the difference in the diagnosis and treatment quality of respiratory diseases in hospitals of different regions and levels, including the allocation of related resources (such as personnel, technology, equipment, information construction, etc.); The status of diagnosis and treatment ability (prevention, diagnosis, treatment, rehabilitation, etc.); Current burden of disease (e.g. morbidity, case fatality rate, average length of stay, average cost of stay, etc.)
3. Promote standardized diagnosis and treatment techniques for major respiratory diseases Relying on the specialized disease collaboration group or innovative unit model, through online and offline academic conferences, continuing medical education, specialized training, visits and exchanges, case discussions, knowledge competitions, wechat public accounts and other new media means, regularly focus on "prevention, diagnosis, treatment, rehabilitation, management, quality control" and many other aspects. Comprehensive and hierarchical precision training and teaching should be carried out to popularize and promote standardized diagnosis and treatment technology schemes for major respiratory diseases, so as to achieve the homogenization of diagnosis and treatment levels for major respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

I. For patients at high risk for VTE 1) Have an expected hospital stay of ≥72 hours for medical and/or surgical treatment II. For patients diagnosed with VTE

1) With clearly diagnosed of deep vein thrombosis or pulmonary thromboembolism

Exclusion Criteria:

I. For patients at high risk for VTE

1. VTE identified on CTPA or lower extremity vein ultrasound at or any time before enrollment
2. Requiring a full dose of anticoagulant treatment before enrollment (e.g., recent VTE, atrial fibrillation).

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: People at high risk of VTE, people diagnosed with VTE
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
A respiratory quality control network platform has been established | 2025.01
  A complete national quality control network platform for the diagnosis and treatment of major respiratory diseases with multi-source data has been built

CONTACTS AND LOCATIONS:
Overall Officials: Zhai Zhenguo, Doctor, Principal Investigator — Department of Respiratory and Critical Care Medicine
Locations (1):
- China-Japanese Friendship Hosptial, Beijing, Beijing Municipality, China